CLINICAL TRIAL: NCT04992325
Title: Anterior Segment- Optical Coherence Tomography as Early Biomarker in Diabetic Retinopathy
Brief Title: AS-OCT Study in Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 2021/07
Record Dates: First submitted 2021-07-25; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes mellitus: The patients with previous diagnosis of type 2 diabetes mellitus, without signs of diabetic retinopathy
  Interventions: Diagnostic Test: Anterior segment-optical coherence tomography
- Healthy subjects: Healthy subjects without actual and previous ocular diseases
  Interventions: Diagnostic Test: Anterior segment-optical coherence tomography

INTERVENTIONS:
Diagnostic Test: Anterior segment-optical coherence tomography — Each subject underwent anterior segment -optical coherence tomography to evaluate the total corneal, epthelium and stromal thicknesses.

SUMMARY:
This study evaluates the corneal features using anterior segment - optical coherence tomography in patients affected by type 2 diabetes mellitus

DETAILED DESCRIPTION:
To investigate the potential role of anterior segment-optical coherence tomography (AS-OCT) in identifying the corneal changes (in particular in total corneal, epithelial and stromal thicknesses) in patients affected by type 2 diabetes mellitus, without signs of diabetic retinopathy at fundus examination.

The AS-OCT could represents a valid early biomarker in these patients.

ELIGIBILITY:
Inclusion Criteria:

* age older than 50 years
* diagnosis of previous type 2 diabetes mellitus
* absence of signs of diabetic retinopathy
* absence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* absence of significant lens opacities, low-quality OCT and OCT-A images

Exclusion Criteria:

* age younger than 50 years
* absence of previous diagnosis of type 2 diabetes mellitus
* presence of signs of diabetic retinopathy
* presence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* presence of significant lens opacities, low-quality OCT and OCT-A images.

Ages: 50 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The participans were older than 50 years with previous diagnosis of type 2 diabetes mellitus without signs of diabetic retinopathy.
  The participans did not present other ophthalmological diseases
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The measurements of corneal features in patients with type 2 diabetes mellitus, using anterior segment-optical coherence tomography | twelve months
  The parameters analyzed by anterior segment-optical coherence tomography angiography were: total corneal, epithelial and stromal thicknesses

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy